CLINICAL TRIAL: NCT06646796
Title: Fibromyalgia: Impact on Pain, Quality of Life of a Complementary Therapy on Primary Health Care
Brief Title: Yoga Impact in Fibromyalgia, Primary Health Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Ines Rosendo, PhD, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 067/2024
Record Dates: First submitted 2024-09-17; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Chronic pain; Yoga; Complementary and alternative medicine
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: In the first phase, the questionnaire will be validated with all patients of the Family Health Unit diagnosed with fibromyalgia who agree to participate. Subsequently, all participants will be asked if they wish to participate in the intervention study, and those who agree will be randomized into either the intervention or control group. The intervention group will engage in Yoga practice with a certified yoga instructor, three times a week for three months. Quality of life scales, a well-being scale, and pain measurement on a numerical scale from 0 to 10 will be applied before and after the intervention, complemented by an open-ended question for qualitative analysis regarding perceived benefits and difficulties.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Group used as comparison.
- Intervention group (Experimental): Yoga practioner group with a certified teacher, 3 times a week during 3 months.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Yoga with certified teacher, 3 times a week during 3 months.
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the effectiveness of a complementary therapy using Yoga within the scope of First Health Care in Portugal, in pain control, quality of life and well-being of the patients with Fibromyalgia. It also, pretends to assess the viability and to identify the barriers to this sort of therapy in the context of Primary Health Care.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic and debilitating pain syndrome characterized by widespread and persistent pain, also affecting sleep quality and cognitive function. It is estimated to affect 3.6% of the population; however, since it is a condition that is often underdiagnosed, the actual numbers may be higher. It is also an incurable disease, so treatment is based on symptom management through pharmacological therapy, which is not always effective. Due to the inadequacy of pharmacological therapy, there is a need for complementary therapies, and despite the limited number of studies conducted in this area, some therapies based on meditative movement (notably yoga) are beginning to emerge, with beneficial effects reported on pain management and quality of life in these patients. Therefore, this study aims to investigate the benefits and feasibility of this type of intervention at the Primary Health Care level.

ELIGIBILITY:
Inclusion Criteria:

* Users of the Family Health Unit diagnosed with Fibromyalgia;
* With cognitive capacity to answer the questionnaire;
* With physical capacity to take part in Yoga classes.

Exclusion Criteria:

* people under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | at the beggining and up to 3 months
  EQ-5D
Pain | at the beggining and up to 3 months
  Visual scale from 0 to 10 to measure pain
Global perception of change | up to 3 months
  Patient Global Impression of Change scale (portuguese validated version)
  1 to 7 (1 is the worst, 7 is the best)

SECONDARY OUTCOMES:
Well-being | at the beggining and up to 3 months
  EADS-21
Benefits perceived | up to 3 months
  Open question answered by the patients trough a written text
Difficulties perceived | up to 3 months
  Open question answered by the patients trough a written text
Replicability and ease of introducing treatment in the context of the Portuguese national health service | up to 3 months
  Open questions and SWOT analysis

CONTACTS AND LOCATIONS:
Locations (1):
- USF Coimbra Centro, Coimbra, Coimbra District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabo-Meseguer A, Cerda-Olmedo G, Trillo-Mata JL. Fibromyalgia: Prevalence, epidemiologic profiles and economic costs. Med Clin (Barc). 2017 Nov 22;149(10):441-448. doi: 10.1016/j.medcli.2017.06.008. Epub 2017 Jul 19. English, Spanish. PMID 28734619
- [Background] Prabhakar A, Kaiser JM, Novitch MB, Cornett EM, Urman RD, Kaye AD. The Role of Complementary and Alternative Medicine Treatments in Fibromyalgia: a Comprehensive Review. Curr Rheumatol Rep. 2019 Mar 4;21(5):14. doi: 10.1007/s11926-019-0814-0. PMID 30830504